CLINICAL TRIAL: NCT00409292
Title: Phase II Study of RAD001 in Previously Treated Patients With Metastatic Pancreatic Cancer
Brief Title: RAD001 in Previously Treated Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Brian Wolpin, MD, MPH, Overall PI, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-197
Record Dates: First submitted 2006-12-06; First posted 2006-12-08 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-07

CONDITIONS: Pancreatic Cancer
Keywords: RAD001; metastatic pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Everolimus

ARMS (1):
- RAD001 (Experimental): RAD001 was administered continuously at a dose of 10 mg daily by mouth until disease progression, unacceptable toxicity, or withdrawal of consent.
  Four weeks of study drug was considered to be one cycle of treatment.
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — Taken orally daily for as long as the participant continues to receive a benefit.

SUMMARY:
The purpose of this research study is to investigate if RAD001 is an effective treatment for pancreatic cancer that has spread and not responded to treatment. Experiments have shown that RAD001 can prevent cells from multiplying. RAD002 has also been tested in laboratory experiments imitating cancer conditions and the results have been promising.

DETAILED DESCRIPTION:
* Participants taking part in this research study will be given a study medication-dosing calendar for each treatment cycle. Each cycle lasts four weeks during which you will be taking the study drug, RAD001, orally every day.
* Participants will come into the clinic every other week during the time of enrollment. At each clinic visit blood work will be taken to monitor the participants health and a physical exam will be performed. CT scans will be repeated every 2 months to assess the tumor.
* Participants will remain on the study as long as they continue to benefit from the study medication.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of pancreatic adenocarcinoma
* 18 years of age or older
* At least one measurable site of disease according to RECIST criteria that has not been previously irradiated. If patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation.
* Treated with gemcitabine-based chemotherapy with documented tumor progression on gemcitabine or intolerance to gemcitabine.
* Prior treatment with no more than 1 prior chemotherapy regimen for metastatic disease.
* Minimum of two weeks since any major surgery, completion of radiation, or completion of all prior systemic anti-cancer therapy.
* ECOG performance status 0-1.
* Life expectancy of greater than 12 weeks.
* Adequate bone marrow and liver function.
* Must be able to swallow tablets.

Exclusion Criteria:

* Prior treatment with an investigational drug within the preceding 4 weeks.
* Prior treatment with an inhibitor of mTOR
* Chronic treatment with systemic steroids or another immunosuppressive agent
* More than one prior chemotherapy treatment for metastatic disease
* Uncontrolled brain or leptomeningeal metastases, including patient who continue to require glucocorticoids for brain or leptomeningeal metastases.
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin
* Patients with chronic renal insufficiency
* Other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study.
* Known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that my significantly alter the absorption of RAD001.
* Active, bleeding diathesis or an oral vitamin K antagonist medication
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Fuchs, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Wolpin BM, Hezel AF, Abrams T, Blaszkowsky LS, Meyerhardt JA, Chan JA, Enzinger PC, Allen B, Clark JW, Ryan DP, Fuchs CS. Oral mTOR inhibitor everolimus in patients with gemcitabine-refractory metastatic pancreatic cancer. J Clin Oncol. 2009 Jan 10;27(2):193-8. doi: 10.1200/JCO.2008.18.9514. Epub 2008 Dec 1. PMID 19047305

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RAD001
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Our study design used a one-stage design with a target accrual of 35 eligible patients, with the assumption that an improvement in PFS at 2 months from 50% to 71% would warrant further study in this patient population.
Arm/Group | RAD001
Number analyzed (Participants) | 33
Age, Customized [Median (Full Range); unit: years] | 61 [39 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: To Assess Progression-free Survival of RAD001 at Two Months in Patients With Metastatic Pancreatic Cancer Whose Disease Has Progressed on Gemcitabine Chemotherapy.
Description: The Outcome Measure is reporting the number of participants experiencing Progression-free Survival at 2 months after treatment.
  The study was designed with a primary end point of progression-free survival (PFS), defined as the time from study entry to documentation of progressive disease or death from any cause. On the basis of prior studies of second-line treatment in metastatic pancreatic cancer, we estimated that such treatment has been associated with a median PFS of 2 months. Our study design used a one-stage design with a target accrual of 35 eligible patients, with the assumption that an improvement in PFS at 2 months from 50% to 71% would warrant further study in this patient population.
Time Frame: two months
Population: On the basis of prior studies of 2nd line treatment in metastatic pancreatic cancer, we estimated a median PFS of 2 months. Our study design used a one-stage design with a target accrual of 35 eligible patients, with the assumption that an improvement in PFS at 2 months from 50% to 71% would warrant further study in this population.
Measure: Number; unit: participants
Groups:
- RAD001: RAD001 was administered continuously at a dose of 10 mg daily by mouth until disease progression, unacceptable toxicity, or withdrawal of consent.
Arm/Group | RAD001
Number analyzed (Participants) | 29
participants | 23
Statistical Analysis 1: Comparison: RAD001; Test type: Superiority or Other; p = 0.10, binomial hypothesis test

2. Secondary Outcome: To Assess the Safety of RAD001 in Patients With Metastatic Pancreatic Cancer
Description: Patients were followed for the duration of their time on treatment and 30 days after their last dose of RAD001. The number of patients with treatment-related adverse events are reported.
Time Frame: Patients were followed for the duration of their time on treatment and 30 days after their last dose of RAD001.
Population: A total of 33 eligible patients received at least 1 week of study drug and are included in our toxicity analyses.
Measure: Number; unit: participants
Arm/Group | RAD001
Number analyzed (Participants) | 33
participants | 33

3. Secondary Outcome: to Assess Response Rate Associated With RAD001 in This Patient Population.
Description: The secondary objectives of the study were to assess tumor response rate and overall survival. Patients were required to have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST). Per RECIST, for target lesions assessed by CT: Complete Response (CR) is Disappearance of all target lesions; Partial Response (PR) is >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) equals CR + PR.
Time Frame: 2 years
Population: Of the 33 patients enrolled, 29 reached restaging. Three patients who did not reach restaging were removed from study because of withdrawal of consent. One patient was removed from study after 8 days of treatment because of worsening of a preexisting perirectal fistula, requiring surgical intervention.
Measure: Number; unit: participants
Arm/Group | RAD001
Number analyzed (Participants) | 29
participants
  Stable Disease as Best Response | 7
  Progressive Disease as Best Response | 22

4. Secondary Outcome: to Assess Overall Survival Associated With RAD001 in This Patient Population.
Description: Overall survival was defined as the time from study entry until death from any cause.
Time Frame: 2 years
Measure: Median (Full Range); unit: months
Groups:
- RAD001: RAD001 was administered continuously at a dose of 10 mg daily by mouth until disease progression, unacceptable toxicity, or withdrawal of consent.
  Four weeks of study drug was considered to be one cycle of treatment.
  RAD001: Taken orally daily for as long as the participant continues to receive a benefit.
Arm/Group | RAD001
Number analyzed (Participants) | 29
months | 4.5 [0.97 to 15.43]

ADVERSE EVENTS:
Arm/Group | RAD001
Serious Adverse Events (participants affected / at risk) | 25/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (N=33)
Lymphocytes (Blood and lymphatic system disorders) | 2
Neutrophils (Blood and lymphatic system disorders) | 3
Platelets (Blood and lymphatic system disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 6
ALT (Hepatobiliary disorders) | 1
Hypercholesterolemia (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Oral Mucositis/Stomatitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (N=33)
Lymphocytes (Blood and lymphatic system disorders) | 8
Neutrophils (Blood and lymphatic system disorders) | 5
Hemoglobin (Blood and lymphatic system disorders) | 17
Platelets (Blood and lymphatic system disorders) | 14
Hypokalemia (Metabolism and nutrition disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 16
ALT (Hepatobiliary disorders) | 3
AST (Hepatobiliary disorders) | 10
Hypercholesterolemia (Metabolism and nutrition disorders) | 6
Fatigue (General disorders) | 16
Nausea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 4
Oral Mucositis/Stomatitis (Gastrointestinal disorders) | 9
Anorexia (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No